CLINICAL TRIAL: NCT03390582
Title: Gut Microbiota is Associated With Autoimmune Thyroid Disease(GD and HT)
Brief Title: Gut Microbiota is Associated With Autoimmune Thyroid Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Yunwei Wei 2017-12-14
Record Dates: First submitted 2017-12-14; First posted 2018-01-04 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2017-12

CONDITIONS: Gut Microbiota
Keywords: Gut Microbiota; Hashimoto Thyroiditis; Graves' Disease; Methimazole; Levothyroxine sodium; 16S rRNA gene; Metabonomics
MeSH Terms: conditions — Hashimoto Disease; Graves Disease | interventions — Methimazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — microbiota DNA are extracted from human feces
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Hashimoto's thyroiditis: Hashimoto's thyroiditis (HT) is an organ-specific autoimmune disease in which both genetic predisposition and environmental factors serve as disease triggers.
- healthy controls: healthy controls are all from normal volunteers
- treatment_naive GD: GD is primarily a humoral disease where autoantibodies are generated against the thyroid stimulating hormone receptor (TSHR) leading to hyperthyroidism.
- treated GD: GD patients treated by Methimazole Pill
  Interventions: Drug: Methimazole Pill

INTERVENTIONS:
Drug: Methimazole Pill — Hyperthyroidism patients are treated with Methimazole Pill according to the guidelines
  Other Names: Methimazole
  Groups: treated GD

SUMMARY:
Autoimmune thyroid disease (AITD), which includes Hashimoto's thyroiditis (HT) and Grave's disease (GD), are the most common organ-specific autoimmune diseases and affect more women than men, with a female-to-male ratio from 5 to 10. Many studies have indicated that alterations in the gut microbiota are important environmental factors in the development of inflammatory and autoimmune diseases. Investigators systematically performed a comparative analysis of the gut microbiota in AITD patients and healthy controls.

DETAILED DESCRIPTION:
Autoimmune thyroid disease (AITD), which includes Hashimoto's thyroiditis (HT) and Grave's disease (GD), are the most common organ-specific autoimmune diseases and affect more women than men, with a female-to-male ratio from 5 to 10. These two diseases are clinically diverse because in HT, T cells aid in the destruction of the thyroid epithelial cells (thyrocytes) and thyroid epithelial structure and eventual fibrous replacement of parenchymal tissue leading to hypothyroidism, whereas GD is primarily a humoral disease where auto-antibodies are generated against the thyroid stimulating hormone receptor (TSHR) leading to hyperthyroidism (2,163-165). However, these diseases still share several immunological features，and the disease may progress from one state to another as the autoimmune process evolves. Many studies have indicated that alterations in the gut microbiota are important environmental factors in the development of inflammatory and autoimmune diseases. Investigators systematically performed a comparative analysis of the gut microbiota in AITD patients and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years
* Male or female gender
* Euthyroidism (normal FT3, FT4, and TSH plasma levels without hormonal therapy)

Exclusion Criteria:

* Pregnancy
* Lactation
* Cigarette smoking
* Alcohol addiction
* Hypertension
* Diabetes mellitus
* Lipid dysregulation
* BMI > 27
* Recent (< 3 months prior) use of antibiotics, probiotics, prebiotics, symbiotics, hormonal medication, proton pump inhibitors, insulin sensitizers or Chinese herbal medicine
* Known history of disease with an autoimmune component such as MS, rheumatoid arthritis, IBS, and IBD
* History of malignancy or any gastrointestinal tract surgery (e.g., gastrectomy, bariatric surgery, colectomy, ileectomy, cholecystectomy or appendectomy).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study Population are aged from 18 to 65 years，which divided into 4 groups:treatment-naive HT, treatment-naive GD, GD treated, healthy controls.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-04-20 (Actual); Primary Completion 2018-12-24 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
16S rRNAgene sequencing was used to measure the diversity of gut microbiota | HC, treatment_naive HT and treatment_naive GD patients samples were collected at the enroll. Treated GD patients were collected until thyroid function resumed to the normal for at least 3 months of methimazole withdrawal
  Intestinal microbes are different in different groups

SECONDARY OUTCOMES:
Thyroid function tested by Chemiluminescence method | Treatment_naive GD and treatment_naive HT patients thyroid function were tested at the enroll and after 3 months
  Serum results are different in different groups and different time point

OTHER OUTCOMES:
Thyroid relative antibody test by Chemiluminescence | Treatment_naive GD and treatment_naive HT patients thyroid function were tested at the enroll and after 3 months
  Serum results are different in different groups and different time point

CONTACTS AND LOCATIONS:
Overall Officials: Wei Yunwei, Study Director — First Affiliated Hospital of Harbin Medical University
Locations (1):
- First affiliated hospital of Harbin medical university, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No